CLINICAL TRIAL: NCT04464577
Title: A Phase 1, Open-label Study to Evaluate the Effect of Fluconazole, Bupropion, or Itraconazole on the Pharmacokinetics and Safety of BMS-986235
Brief Title: A Study to Evaluate the Effect of Fluconazole, Bupropion, or Itraconazole on the Drug Levels and Safety of BMS-986235
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed.
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CV018-014
Record Dates: First submitted 2020-03-23; First posted 2020-07-09 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Healthy Participants
MeSH Terms: interventions — Fluconazole; Bupropion; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: BMS-986235+Fluconazole (Experimental)
  Interventions: Drug: Fluconazole; Drug: BMS-986235
- Arm B: BMS-986235+ Bupropion (Experimental)
  Interventions: Drug: Bupropion; Drug: BMS-986235
- Arm C: BMS-986235+ Itraconazole (Experimental)
  Interventions: Drug: Itraconazole; Drug: BMS-986235

INTERVENTIONS:
Drug: Fluconazole — Specified Dose on Specified Days
  Arms: Arm A: BMS-986235+Fluconazole
Drug: Bupropion — Specified Dose on Specified Days
  Arms: Arm B: BMS-986235+ Bupropion
Drug: Itraconazole — Specified Dose on Specified Days
  Arms: Arm C: BMS-986235+ Itraconazole
Drug: BMS-986235 — Specified Dose on Specified Days

SUMMARY:
This study will evaluate the effect of inhibitors, at steady state, on the drug levels, safety, and tolerability of BMS-986235 when taken by healthy participants. The inhibitors to be utilized in this study are fluconazole, bupropion, and itraconazole.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 18.0 kg/m2 to 32.0 kg/m2, inclusive, at screening.
* Males and females must agree to follow specific methods of contraception, if applicable.
* Healthy participants, as determined by no clinically significant deviation from normal in physical examination, ECGs, and clinical laboratory determinations, and no significant findings in medical history.

Exclusion Criteria:

* Women of childbearing potential (WOCBP), women who are pregnant or breastfeeding
* Inability to tolerate oral medication
* Known previous exposure to BMS-986235.

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2021-06-07 (Estimated); Study Completion 2021-06-08 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUC(0-T)) of BMS-986235 with fluconazole | Day 12
Maximum plasma concentration (Cmax) of BMS-986235 with fluconazole | Day 12
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC(INF)) of BMS-986235 with fluconazole | Day 12
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC(INF)) of BMS-986235 with bupropion | Day 13
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUC(0-T)) of BMS-986235 with bupropion | Day 13
Maximum plasma concentration (Cmax) of BMS-986235 with bupropion | Day 13
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUC(0-T)) of BMS-986235 with itraconazole | Day 9
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC(INF)) of BMS-986235 with itraconazole | Day 9
Maximum plasma concentration (Cmax) of BMS-986235 with itraconazole | Day 9
Area under the plasma concentration-time curve from time 0 extrapolated to infinity (AUC(INF)) of BMS-986235 | Day 1
Area under the plasma concentration-time curve from time 0 to time of last quantifiable concentration (AUC(0-T)) of BMS-986235 | Day 1
Maximum plasma concentration (Cmax) of BMS-986235 | Day 1

SECONDARY OUTCOMES:
Incidence of Nonserious Adverse Events (AEs) | Up to 49 days
Incidence of Serious Adverse Events (SAEs) | Up to 77 days
Incidence of AEs leading to discontinuation | Up to 16 days
Number of clinically significant changes from baseline in vital signs: Body Temperature | Up to 44 days
Number of clinically significant changes from baseline in physical examinations | Up to 44 days
Number of clinically significant changes in clinical laboratory tests: Hematology | Up to 44 days
Number of clinically significant changes in clinical laboratory tests: Clinical Chemistry | Up to 44 days
Number of clinically significant changes in clinical laboratory tests: Coagulation | Up to 44 days
Number of clinically significant changes in clinical laboratory tests: Urinalysis | Up to 44 days
Number of clinically significant changes from baseline in vital signs: Respiratory Rate | Up to 44 days
Number of clinically significant changes from baseline in vital signs: Heart Rate | Up to 44 days
Number of clinically significant changes from baseline in vital signs:Blood Pressure | Up to 44 days
Number of clinically significant changes in electrocardiogram (ECG) | Up to 44 days
Number of clinically significant changes in vital signs: Oxygen saturation (the amount of oxygen in blood (SpO2)) | Up to 44 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution, Lenexa, Kansas
  - Local Institution, Salt Lake City, Utah

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm